CLINICAL TRIAL: NCT04200755
Title: A Randomized, Placebo-controlled Phase IIa Clinical Trial to Evaluate the Efficacy and Safety of Subcutaneous Dupilumab in Localized Scleroderma
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of Dupilumab in Localized Scleroderma
Acronym: DupiMorph
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Sabine Eming, Principal Coordinating Investigator, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Uni-Koeln-3815; 2019-002036-90 (EudraCT Number)
Record Dates: First submitted 2019-12-10; First posted 2019-12-16 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Localized Scleroderma
Keywords: Morphea
MeSH Terms: conditions — Scleroderma, Localized | interventions — dupilumab; Solutions; Injections

STUDY DESIGN:
Intervention Model Description: Randomized, multi-center, double-blind, placebo controlled, parallel group, multiple dose, phase IIa trial
Who Masked: Participant, Investigator
Masking Description: Permuted blocks of varying length with allocation ratio (verum:placebo = 2:1); double-blind, i.e. patients and investigators are masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dupilumab (Experimental): 30 patients; Dupilumab s.c. injection; 2 ready-to-use syringes (600 mg) initial (V1), 1 ready-to-use syringe (300 mg) every 14 days (V2- V13) Dupilumab s.c. injection in healthy skin, 24 weeks
  Interventions: Drug: Dupilumab 300Mg Solution for Injection
- Placebo (Placebo Comparator): 15 patients; placebo s.c. injection; 2 ready-to-use syringes initial (V1), 1 ready-to-use syringe every 14 days (V2-V13) placebo s.c. injection in healthy skin, 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dupilumab 300Mg Solution for Injection — First dose: 600 mg (2 syringes); subsequent doses: 300 mg (1 syringe)
  Other Names: Dupixent
  Arms: Dupilumab
Other: Placebo — First dose: 2 syringes, no active substance; subsequent doses: 1 syringe, no active substance
  Arms: Placebo

SUMMARY:
The DupiMorph study evaluates the efficacy of Dupilumab in localized scleroderma patients. Dupilumab is approved in the US and EU for the treatment of moderate/severe atopic dermatitis and since 2018 in the US for severe asthma therapy.

DETAILED DESCRIPTION:
Localized scleroderma (LS) comprises a heterogenous group of sclerotic skin disorders. The incidence of LS is reported to be approximately 27 cases/ 1x106 and is hence approximately 2-3-fold higher compared to systemic scleroderma. Although in most cases not lethal the disease can significantly impact quality of life. Depending on the location of fibrosis, the disorder can cause bone deformities, alopecia, skin atrophy or lesions with severe hypo-/hyperpigmentation.

The disease is pathomechanistically poorly understood and no effective therapy is currently approved. The most promising treatments up to date include methotrexate ± pulsed corticosteroids or phototherapy with PUVA or UVA1. Yet, the number of treated patients in these studies is low. The response rates are low and inconsistent with approximately 50% of patients treated with UVA1 experience a recurrence within three years. There are no studies on efficacy of topical corticosteroids in LS. Small pilot studies and few case reports describe regression of lesions after topical calcineurin inhibitors. In addition, current therapies can only be applied for a short time during the acute phase due to the side effect profile after long-term use (e.g. skin atrophy in response to topical steroids, skin cancer in response to long term UV therapy, multiple side effects by long- term use of methotrexate and/or corticosteroids). Hence, this study evaluates, in comparison with placebo, the efficacy of Dupilumab administered subcutaneously every 14 days in patients with Morphea (plaque type) or generalized localized scleroderma (affecting at least three anatomic sites).

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or female ≥18 years of age on the day the study informed consent is signed
* Out-patient status
* Caucasian
* Morphea (plaque type) or Generalized localized scleroderma (affecting at least three anatomic sites)
* At least one lesions with lilac ring (active phase of the disease);
* Activity of LS within the last 12 month (as defined by progression of size or new developing plaque)
* For women of childbearing potential: negative pregnancy test at Visit 1
* For women of childbearing potential: Use of effective method of contraception from 4 weeks prior to enrolment, throughout study treatment until 12 weeks after the last IMP dose.
* Written informed consent signed

Exclusion Criteria:

* Systemic immunosuppressive therapy or UV therapy less than 3 months before enrollment.
* Participation in another trial of IMPs or devices parallel to, or less than 6 months before or previous participation in this trial
* Pregnancy or breastfeeding mother
* Diagnosis of other significant chronic inflammatory or autoimmune disorders. Patients with the following autoimmune disorders are excluded from the study: Multiple sclerosis, primary biliary cirrhosis, type I diabetes mellitus. Patients with the following autoimmune disorders are regarded as eligible: Lichen sclerosus, vitiligo, alopecia arthritis, thyroid diseases (e.g. Hashimoto disease). Patients with any autoimmune disorder not listed above should only be included after consultation with the principal coordinating investigator.
* Topical immunosuppressive therapy less than 1 month before enrollment
* Concurrent phototherapy
* Known infection with helminths (helminthosis)
* Any condition or laboratory abnormality that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study or may interfere with the assessments included in the study. E.g. uncontrolled psychiatric illness or history of clinical relevant drug abuse.
* Known hypersensitivity to any components of the IMP
* Treatment with a live (attenuated) vaccine within 3 months prior to enrollment
* History of malignancy (except patients with completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin)
* Known diagnosis of active tuberculosis or non-tuberculous mycobacterial infection or latent untreated tuberculosis unless it is well documented by a specialist that the patient has been adequately treated
* Known diagnosis of HIV, HBV or HCV infection
* Regular use (more than 2 visits per week) of a tanning booth/parlor
* Known diagnosis of asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
LoSCAT target lesion | Baseline to End of Treatment Visit, 24 weeks
  Treatment response is assessed using the LoSCAT (Localized Scleroderma Cutaneous Assessment Tool). Target lesion will be assessed at Baseline and End of Treatment. Score reduction by 50% after 24 weeks (End of Treatment Visit V14) compared to Baseline Visit (V1) is defined as treatment response.

SECONDARY OUTCOMES:
mLoSSI all lesions | Baseline to Follow-Up Visit, 48 weeks
  Change in mLoSSI (Localized Scleroderma Skin Activity Index) of all existing lesions during treatment, at End of Treatment Visit and during follow-up
LoSDI all lesions | Baseline to Follow-Up Visit, 48 weeks
  Change in LoSDI (Localized Scleroderma Skin Damage Index) of all existing lesions during treatment, at End of Treatment Visit and during follow-up
Number of lesions | Baseline to Follow-Up Visit, 48 weeks
  Count of all existing non-target and new lesions on the entire integument during treatment, at End of Treatment Visit and during follow-up
DLQI | Baseline to Follow-Up Visit, 48 weeks
  Change in DermatoLogy Quality of life Index (DLQI). The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
RNAseq | Baseline to End of Treatment Visit, 24 weeks
  Gene signature of localized scleroderma after Dupilumab treatment: RNA- seq of tissue biopsies obtained from the lesion (lilac ring, optional: center) before (baseline visit V1) and after treatment (EoT V14) and healthy skin before treatment
RT-qPCR | Baseline to End of Treatment Visit, 24 weeks
  Quantification of change in gene expression of genes identified by RNAseq in tissue of localized scleroderma patients after Dupilumab treatment: RT-qPCR of tissue biopsies obtained from the lesion (lilac ring, optional: center) before (baseline visit V1) and after treatment (End of Treatment Visit V14) and healthy skin before treatment
Adverse events (AEs) | Baseline to Follow-Up Visit, 48 weeks
  Adverse events will be documented throughout the study
Physical examination | Baseline to Follow-Up Visit, 48 weeks
  Physical examination (general appearance including skin, head and throat (head, eyes, ears, nose, and throat), lymph nodes, respiratory, cardiovascular, musculoskeletal, and neurological systems) will be documented throughout the study.
Body weight | Baseline to Follow-Up Visit, 48 weeks
  Body weight will be documented throughout the study.
Blood pressure | Baseline to Follow-Up Visit, 48 weeks
  Blood pressure will be documented throughout the study.
Pulse rate | Baseline to Follow-Up Visit, 48 weeks
  Pulse rate will be documented throughout the study.
Body temperature | Baseline to Follow-Up Visit, 48 weeks
  Body temperature will be documented throughout the study.
Haematocrit (HcT) | Baseline to Follow-Up Visit, 48 weeks
  Haematocrit (HcT) will be documented at End of Treatment Visit and during follow-up
Haemoglobin | Baseline to Follow-Up Visit, 48 weeks
  Haemoglobin (Hgb) will be documented at End of Treatment Visit and during follow-up
Blood cell count | Baseline to Follow-Up Visit, 48 weeks
  Platelet count and differential White blood cell count will be documented at End of Treatment Visit and during follow-up
Blood Enzymes | Baseline to Follow-Up Visit, 48 weeks
  Clinical Chemistry parameters (Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Gamma-glutamyl transferase (GGT), Lactic dehydrogenase (LDH)) will be documented at End of Treatment Visit and during follow-up
Clinical Chemistry | Baseline to Follow-Up Visit, 48 weeks
  Clinical Chemistry parameters (Creatinine) will be documented at End of Treatment Visit and during follow-up
Anti-nuclear antibodies (ANAs) levels | Baseline to Follow-Up Visit, 48 weeks
  Change in anti-nuclear antibodies (ANAs) levels
Serum cytokine levels | Baseline to Follow-Up Visit, 48 weeks
  Change in serum levels of IL-4, IL-5, IL-13, periostin, dipeptidyl peptidase-4

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Eming, Prof. Dr., Principal Investigator — University of Cologne
Locations (4):
- Germany (4):
  - Charité - Universitätsmedizin Berlin Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Uniklinik Köln, Klinik für Dermatologie und Venerologie, Cologne
  - Helios St. Elisabeth Klinik Oberhausen, Klinik für Dermatologie, Venerologie und Allergologie, Oberhausen
  - Universitäts-Hautklinik Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No